CLINICAL TRIAL: NCT00358384
Title: A Study to Investigate the Irritation Potential on Healthy Intact Skin and Effect on Psoriatic Skin of Topical Applications of GW786034
Brief Title: Chronic Plaque Psoriasis Study With Topical Formulation Of GW786034
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: RES104031
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Psoriasis
Keywords: tolerability; safety; angiogenesis; vascular endothelial growth factor; pharmacodynamics; pharmacokinetics; microplaque; VEGF; GW786034
MeSH Terms: conditions — Psoriasis | interventions — pazopanib; Betamethasone Valerate; calcipotriene

ARMS (6):
- Subjects receiving treatment A (Experimental): Eligible subjects will receive 0.1 percent pazopanib ointment.
  Interventions: Drug: Pazopanib
- Subjects receiving treatment B (Experimental): Eligible subjects will receive 0.5 percent pazopanib ointment.
  Interventions: Drug: Pazopanib
- Subjects receiving treatment C (Experimental): Eligible subjects will receive 1 percent pazopanib ointment.
  Interventions: Drug: Pazopanib
- Subjects receiving treatment D (Placebo Comparator): Eligible subjects will receive pazopanib vehicle as negative control.
  Interventions: Drug: Pazopanib vehicle
- Subjects receiving treatment E (Placebo Comparator): Eligible subjects will receive 0.1 percent betamethasone valerate ointment as steroid positive control.
  Interventions: Drug: Betamethasone valerate
- Subjects receiving treatment F (Placebo Comparator): Eligible subjects will receive 0.005 percent calcipotriol ointment as vitamin D agonist positive control.
  Interventions: Drug: Calcipotriol

INTERVENTIONS:
Drug: Pazopanib — Pazopanib will be available in dosing strengths of 0.1, 0.5 and 1 percent.
  Arms: Subjects receiving treatment A; Subjects receiving treatment B; Subjects receiving treatment C
Drug: Pazopanib vehicle — Pazopanib vehicle will be given to subjects.
  Arms: Subjects receiving treatment D
Drug: Betamethasone valerate — Betamethasone valerate ointment with 0.1 percent concentration will be given to subjects.
  Arms: Subjects receiving treatment E
Drug: Calcipotriol — Calcipotriol ointment with 0.005 percent concentration will be given to subjects.
  Arms: Subjects receiving treatment F

SUMMARY:
This study is an exploratory study to evaluate the effectiveness, safety and tolerability of three concentrations of GW786034 ointment following treatment to small areas of stable psoriatic plaques. Dosing will proceed using a microplaque approach, where small volumes of ointment will be applied under full occlusion to representative psoriatic plaques. The effectiveness of topical GW786034 treatments and controls will be explored using visual intensity assessments in addition to dermal imaging and histological surrogates of disease activity.

ELIGIBILITY:
Inclusion criteria:

* Stable (2-3 months) chronic plaque psoriasis covering greater than 5% body surface area (as determined by PASI palm method).
* Other than having chronic plaque psoriasis, subject is health and ambulatory.
* Women will be eligible to enter the study if they are of non-child-bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile).
* Must have at least two clinically similar lesions with the following characteristics as deemed by the dermatologist: Moderate to severe in elevation (thickness), erythema, and scaling (with a total score of at least 6 for each target lesion, when assessed using a 0-4 PASI score). Located on the trunk, buttocks, thighs or upper arms. Are of a sufficient size that will allow the application of three occlusive patches.

Exclusion criteria:

* Guttate, erythrodermic, or pustular psoriasis.
* Psoriasis is spontaneously improving.
* Have had psoriasis that was unresponsive to adequately dosed (> 10 weeks) cyclosporine.
* Any systemic disorder or active skin disease (other than psoriasis) or subjects who present with scars, moles, tattoos, body piercings, sunburn in the test area.
* History of congestive heart failure (NYHA Class 3 or 4), myocardial infarction, coronary artery bypass graft, percutaneous transluminal balloon angioplasty, cerebrovascular accident, chronic or intermittent oedema.
* Blood pressure of greater than 150mmHg systolic and /or 95mmHg diastolic following triplicate measurements taken 5 minutes apart.
* Presence of unstable or severe angina or coronary insufficiency.
* Uncontrolled bacterial, viral, or fungal infection.
* Congenital or acquired immunodeficiency.
* History of malignancy within the last five years, except for surgically cured skin carcinoma or cervical dysplasia (CIN I-II).
* An unwillingness of male subjects to use a condom/spermicide in addition to having their female partner use another form of contraception if the woman could become pregnant from the time of the first dose of study medication until 5 half-lives of the drug have elapsed following removal of the last dose of study medication.
* An unwillingness of male subjects to abstain from sexual intercourse with pregnant or lactating women from the time of first dose of study medication until five half-lives or 5 days (whichever is longer) following removal of the last dose of study medication.
* Prolonged exposure to the sun (or tanning beds) during the study.
* Systemic anti-psoriasis therapy, including but not limited to: acitretin, cyclosporine, isotretinoin, infliximab, entercept, alefacept, oral steroids and psoralen during the 4 weeks prior to the first dose of study medication and throughout the study.
* Concomitant use of phototherapy or photochemotherapy.
* Concomitant use of lithium, antimalarials, interferons.
* Systemic beta-blockers are permitted provided the dose is stable for four weeks before baseline and remains stable throughout the study.
* Concomitant use of anti-arthritis therapies with known propensity for hepatotoxicity (i.e. diclofenac, gold, D-penicillamine, leflunomide).
* Use of topical or intralesional treatments for psoriasis (e.g. mid- or high-potency topical corticosteroids) within 2 weeks prior to Day 1 and throughout the study, except for class VI or VII topical steroid treatments (Desonide, or 2.5% hydrocortisone) which will be allowed on the face.
* Concomitant use of non-drug therapies (i.e. herbal products or alternative therapies) for psoriasis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-09-26 (Actual); Primary Completion 2006-02-24 (Actual); Study Completion 2006-02-24 (Actual)

PRIMARY OUTCOMES:
Visual assessment and clinical scoring of lesion treatment areas using modified Psoriasis Area Scoring Index (PASI) target lesion assessment scale Clinical lab tests vital signs adverse events clinical monitoring/observation | Up to 8 weeks

SECONDARY OUTCOMES:
Laser doppler imaging,epidermal thickness by histology skin biopsies Primary pharmacokinetic endpoints AUC(0-t) and Cmax of GW786034 in plasma following repeat dosing | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Paris, France

REFERENCES:
- See also: Results for study RES104031 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/RES104031?search=study&study_ids=RES104031#rs